CLINICAL TRIAL: NCT04597307
Title: IN.PACT™ Quality of Life Post-Reimbursement Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: IN.PACT™ QoL PSR
Record Dates: First submitted 2020-09-16; First posted 2020-10-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Disease; Atherosclerosis of Femoral Artery; Atherosclerosis of Popliteal Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- IN.PACT™ Admiral™ DCB Cohort: De novo patients not previously treated with a DCB who are successfully treated with the IN.PACT™ Admiral™ DCB (ability to cross the target lesion).
  Interventions: Combination Product: IN.PACT™ Admiral™ Drug Coated Balloon (DCB)

INTERVENTIONS:
Combination Product: IN.PACT™ Admiral™ Drug Coated Balloon (DCB) — For percutaneous transluminal angioplasty (PTA) in subjects with obstructive disease of the peripheral arteries.

SUMMARY:
To prospectively collect and assess the perception of health-related Quality of Life, Pain and Walking Ability.

DETAILED DESCRIPTION:
To provide both the French National Authority for Health and the French Economic Committee for Health Products requested information on patient-reported outcomes for the IN.PACT™ Admiral™ Drug-Coated Balloon. Patients will be followed using routine clinical practice and the collection of two validated instruments: EuroQOL EQ-5D Quality of Life questionnaire and the Walking Impairment Questionnaire (WIQ).

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible product
* Patient is consented within the enrollment window of the treatment/therapy received

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results (i.e. no required intervention that could affect interpretation of all-around product safety and or effectiveness)

Note: For this study, de novo patients will be enrolled to assess EQ-5D and WIQ at baseline and follow-up. Patients cannot be treated in the same procedure with a competitor drug-coated (DCB) or drug-eluting (DES) in the vessel segment treated with IN.PACT Admiral.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with obstructive disease of the peripheral arteries that will have a percutaneous transluminal angioplasty (PTA) with the IN.PACT™ Admiral™ Drug Coated Balloon (DCB).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life EQ-5D-5L French Index Score Change | Baseline & 12 months after endovascular procedure
  Primary Objective: Assess the mean change of patient reported outcomes between pre-procedure visit (baseline) and 12 months after the endovascular procedure of the EQ-5D-5L Questionnaire using the French Index Score (from -0.530 to 1.000 with 1 being better) in the treatment of de novo PTA subjects with obstructive disease of peripheral arteries with the IN.PACT™ Admiral™ DCB.
Walking Ability Change | Baseline & 12 months after endovascular procedure
  Primary Objective: Assess the mean change of patient reported outcomes between pre-procedure visit (baseline) and 12 months after the endovascular procedure of the Walking Impairment Questionnaire (WIQ) (0 to 100% with 100% being better) in the treatment of de novo PTA subjects with obstructive disease of peripheral arteries with the IN.PACT™ Admiral™ DCB.

SECONDARY OUTCOMES:
Quality of Life EQ-5D-5L French Index Score Change Over Time | Baseline, 30 days, 12 months and 24 months from the endovascular procedure
  Assess the mean change of patient reported outcomes over time of EQ-5D-5L French Index Score (from -0.530 to 1.000 with 1 being better) collected at pre-procedure visit (baseline) and at 30 days, 12 months, and 24 months from the endovascular procedure in de novo patients treated with the IN.PACT™ Admiral™ DCB.
  In addition, the EQ-5D VAS Score (0 to 100 with 100 being better) will be assessed using the mean change between pre-procedure visit (baseline) and 12 months after endovascular procedure as well as the mean change over time collected at preprocedure visit (baseline) and at 30 days, 12 months, and 24 months from the endovascular procedure with the IN.PACT™ Admiral™ DCB.
Walking Ability Change Over Time | Baseline, 30 days, 12 months and 24 months from the endovascular procedure
  Assess the mean change of patient reported outcomes over time of the WIQ composite score (0 to 100% with 100% being better) collected at pre-procedure visit (baseline) and at 30 days, 12 months, and 24 months from the endovascular procedure in de novo patients treated with the IN.PACT™ Admiral™ DCB.
  In addition, the WIQ questions for Walking Impairment, Walking Distance, Walking Speed, and Stair Climbing will be assessed using the mean change between pre-procedure visit (baseline) and 12 months after endovascular procedure as well as the mean change over time collected at preprocedure visit (baseline) and at 30 days, 12 months, and 24 months from the endovascular procedure with the IN.PACT™ Admiral™ DCB.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Yann Goueffic, MD, PhD, Principal Investigator — Hôpital Paris St Joseph
Locations (9):
- France (9):
  - Hopitaux Universitaires Paris lle-France Ouest- Hopital Ambroise- Pare, Boulogne
  - CHRU Brest Cavale Blanche, Brest
  - Centre Hospitalier Clermont-Ferrand-Gabriel-Montpied, Clermont-Ferrand
  - Groupe hospitalier Paris Saint-Joseph, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - CHU de Rennes, Rennes
  - Clinique Rhena, Strasbourg
  - Hopitaux Universitaires de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No